CLINICAL TRIAL: NCT02727517
Title: Early or Late Cord Clamping in the Depressed Neonate - a Randomized Controlled Study in a Low-income Facility Setting for Improved Early Neonatal Outcome
Brief Title: Early or Late Cord Clamping in the Depressed Neonate
Acronym: NepCordIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: UNICEF (Other); Ministry of Health and Population, Nepal (Other Government); Swedish Society for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NEPRESUSC16
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Neonatal Disorder; Asphyxia Neonatorum
Keywords: Resuscitation; Cord clamping
MeSH Terms: conditions — Infant, Newborn, Diseases; Asphyxia Neonatorum | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early (≤ 60 seconds) cord clamping (Active Comparator): Early (≤ 60 seconds) cord clamping
  Interventions: Procedure: Early (≤ 60 seconds) cord clamping
- Delayed cord clamping (Active Comparator): Delayed (≥ 180 seconds) cord clamping
  Interventions: Procedure: Delayed (≥ 180 seconds) cord clamping

INTERVENTIONS:
Procedure: Early (≤ 60 seconds) cord clamping — If the infant don't breathe, the umbilical cord is clamped (≤ 60 seconds) and cut and resuscitation will be provided at a resuscitation table
  Other Names: Immediate clamping
  Arms: Early (≤ 60 seconds) cord clamping
Procedure: Delayed (≥ 180 seconds) cord clamping — If the infant don't breathe, the umbilical cord is not clamped and cut until after 180 seconds. Initial resuscitation will be provided bedside to the mother
  Other Names: Late cord clamping; Deferred cord clamping; Optimal cord clamping
  Arms: Delayed cord clamping

SUMMARY:
This study evaluates the hypothesis that delayed compared to early umbilical cord clamping will improve neonatal transition in terms of circulation and breathing during resuscitation.

DETAILED DESCRIPTION:
At the time of birth, the infant is still attached to the placenta via the umbilical cord. The infant is usually separated from the placenta by clamping the cord with two clamps. Early cord clamping has been generally advised to be carried out in the first 30 seconds after birth, regardless of whether the cord pulsation has ceased. However, arguments against early cord clamping include the reduction in the amount of placental transfusion and any associated benefits of extra blood volume, as delayed clamping allows time for a transfer of the fetal blood in the placenta to the infant at the time of birth.

The study will evaluate the effect of early versus delayed cord clamping in a low-income setting in children that do not spontaneously start to breathe. The randomized controlled trial will be carried out at Paropakar Maternity and Women's Hospital (PMWH) in Kathmandu.

The trial will fill several important gaps in relation to early and delayed cord clamping and results.

ELIGIBILITY:
Inclusion Criteria:

* Newborn in need of resuscitation measures (no or irregular breathing despite thorough drying and additional stimulation within one minute after birth)
* Gestational age ≥ 33 weeks

Exclusion Criteria:

Monochorionic twins (from an ultrasound scan) or clinical evidence of twin-twin transfusion syndrome, triplets or higher order multiple pregnancy, and fetuses with known congenital malformation

Ages: 33 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Blood oxygen saturation | 10 minutes after birth
  Measured with a pulse oximeter

SECONDARY OUTCOMES:
Blood oxygen saturation | 5 minutes after birth
  Measured with a pulse oximeter
Timing of reaching > 90 % in oxygen saturation | Within 10 minutes after birth
  Measured with a pulse oximeter
Newborn heart rate | At 1 minute after birth
  Measured with a pulse oximeter (preferred), fetal heart monitor or manually
Newborn heart rate | At 5 minutes after birth
  Measured with a pulse oximeter (preferred), fetal heart monitor or manually
Newborn heart rate | At 10 minutes after birth
  Measured with a pulse oximeter (preferred), fetal heart monitor or manually
Apgar score | At 1 minute after birth
  Assessed by staff, composite of heart rate, breathing effort, skin color, muscle tone and reflexes
Apgar score | At 5 minutes after birth
  Assessed by staff, composite of heart rate, breathing effort, skin color, muscle tone and reflexes
Apgar score | At 10 minutes after birth
  Assessed by staff, composite of heart rate, breathing effort, skin color, muscle tone and reflexes
Pulsatility index | At 5 minutes after birth
  Measured with a pulse oximeter
Pulsatility index | At 10 minutes after birth
  Measured with a pulse oximeter
Timing of establishing spontaneous breathing | Within 10 minutes after birth
  Assessed by staff present
Timing of first cry | Within 10 minutes after birth
  Assessed by staff present
Timing of moving baby from mother to resuscitation table (if applicable | Within 10 minutes after birth
  Assessed by staff present
Rectal temperature | At 30 minutes after birth
  Assessed by staff present

OTHER OUTCOMES:
Presence at one day of age | 24 hours
  The place of stay for newborn at one day of age

CONTACTS AND LOCATIONS:
Overall Officials: Ashish KC, MD PhD, Principal Investigator — Uppsala University; Ola Andersson, MD PhD, Principal Investigator — Uppsala University
Locations (1):
- Paropakar Maternity and Women's Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niermeyer S, Velaphi S. Promoting physiologic transition at birth: re-examining resuscitation and the timing of cord clamping. Semin Fetal Neonatal Med. 2013 Dec;18(6):385-92. doi: 10.1016/j.siny.2013.08.008. Epub 2013 Sep 19. PMID 24055300
- [Derived] Xodo S, Xodo L, Baccarini G, Driul L, Londero AP. Does Delayed Cord Clamping Improve Long-Term (>/=4 Months) Neurodevelopment in Term Babies? A Systematic Review and a Meta-Analysis of Randomized Clinical Trials. Front Pediatr. 2021 Apr 12;9:651410. doi: 10.3389/fped.2021.651410. eCollection 2021. PMID 33912524
- [Derived] Andersson O, Rana N, Ewald U, Malqvist M, Stripple G, Basnet O, Subedi K, Kc A. Intact cord resuscitation versus early cord clamping in the treatment of depressed newborn infants during the first 10 minutes of birth (Nepcord III) - a randomized clinical trial. Matern Health Neonatol Perinatol. 2019 Aug 29;5:15. doi: 10.1186/s40748-019-0110-z. eCollection 2019. PMID 31485335